CLINICAL TRIAL: NCT02646748
Title: A Platform Study Exploring the Safety, Tolerability, Effect on the Tumor Microenvironment, and Efficacy of Pembrolizumab + INCB Combinations in Advanced Solid Tumors
Brief Title: Pembrolizumab Combined With Itacitinib (INCB039110) and/or Pembrolizumab Combined With INCB050465 in Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 39110-107
Record Dates: First submitted 2016-01-04; First posted 2016-01-06 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Colorectal Cancer (CRC); Endometrial Cancer; Melanoma; Head and Neck Cancer; Lung Cancer; MMR-deficient Tumors; Breast Cancer; Pancreatic Cancer; Renal Cell Carcinoma (RCC); Solid Tumors; UC (Urothelial Cancer)
Keywords: Advanced
MeSH Terms: conditions — Colorectal Neoplasms; Endometrial Neoplasms; Melanoma; Head and Neck Neoplasms; Lung Neoplasms; Breast Neoplasms; Pancreatic Neoplasms; Carcinoma, Renal Cell | interventions — pembrolizumab; itacitinib; INCB039110; parsaclisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- pembrolizumab + itacitinib (Experimental): Part 1a Group A will utilize an open-label 3+3 dose-escalation design based on observing each dose level for a period of 21 days.
  Part 1b Group A-1 and Group A-2 will evaluate the MTD or PAD of itacitinib in combination with pembrolizumab in subjects with select solid tumors.
  Interventions: Drug: Pembrolizumab; Drug: itacitinib
- pembrolizumab + INCB050465 (Experimental): Part 1a Group B will utilize an open-label 3+3 dose-escalation design based on observing each dose level for a period of 21 days.
  Part 1b Group B-1 and Group B-2 will evaluate the MTD or PAD of INCB050465 in combination with pembrolizumab in subjects with select solid tumors.
  Part 2 will evaluate the combination of INCB050465 in combination with pembrolizumab in subjects with small cell lung cancer, non-small lung cancer and urothelial cancer.
  Interventions: Drug: Pembrolizumab; Drug: INCB050465

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg IV Q3W.
Drug: itacitinib — Itacitinib tablets administered orally once daily.
  Other Names: INCB039110
  Arms: pembrolizumab + itacitinib
Drug: INCB050465 — INCB050465 tablets administered orally once daily.
  Arms: pembrolizumab + INCB050465

SUMMARY:
This is an open-label, multicenter, Phase 1b platform study in subjects with advanced or metastatic solid tumors (Part 1a) and subjects with selected solid tumors (Part 1b and Part 2). Two treatment groups (Group A and Group B) will be evaluated

Part 1a utilizes a 3+3 design to evaluate pembrolizumab and INCB combinations in advanced solid tumors. Group A will evaluate a JAK inhibitor with JAK1 selectivity itacitinib (INCB039110) in combination with pembrolizumab (MK-3475) and Group B will evaluate a PI3K-delta inhibitor (INCB050465) in combination with pembrolizumab to determine the maximum tolerated dose (MTD) or PAD and recommend a dose for the Part 1b safety expansion with each combination.

Once the recommended dose has been identified in Part 1a, subjects with select solid tumor types will be enrolled into safety expansion cohorts based upon prior treatment history with a PD-1 pathway-targeted agent (Part 1b) for each combination.

Part 2 utilizes a Simon 2-Stage design to evaluate INCB050465 in combination with pembrolizumab in patients with small cell lung cancer (SCLC) and a 1 stage design to evaluate the combination in patients with non-small cell lung cancer (NSCLC) and urothelial cancer (UC).

DETAILED DESCRIPTION:
This is an open-label, Phase 1b, 3 Part (Part 1a, Part 1b, and Part 2), multi-center study.

Part 1a utilizes a 3+3 design to evaluate pembrolizumab and INCB combinations in advanced solid tumors. Group A will evaluate a JAK inhibitor with JAK1 selectivity itacitinib (INCB039110) in combination with pembrolizumab (MK-3475) and Group B will evaluate a PI3K-delta inhibitor (INCB050465) in combination with pembrolizumab to determine the maximum tolerated dose (MTD) or PAD and recommend a dose for the Part 1b safety expansion with each combination.

Once the recommended dose has been identified in Part 1a, subjects with endometrial cancer, gastric cancer, melanoma, microsatellite unstable (MSI) colorectal cancer or other MMR-deficient tumors, non-small cell lung cancer, renal cell carcinoma, head and neck squamous cell carcinoma, triple negative breast cancer, pancreatic ductal carcinoma, or transitional cell carcinoma of the genitourinary tract will be enrolled into safety expansion cohorts based upon prior treatment history with a PD-1 pathway-targeted agent (Part 1b) for each combination.

Part 2 utilizes a Simon 2-Stage design to evaluate INCB050465 in combination with pembrolizumab in patients with small cell lung cancer (SCLC) and a 1 stage design to evaluate the combination in patients with non-small cell lung cancer (NSCLC) and urothelial cancer (UC).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 years or older.
* Willingness to provide written informed consent for the study.
* Has a core or excisional baseline tumor biopsy specimen available or willingness to undergo a pre study treatment tumor biopsy to obtain the specimen.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Presence of measureable disease based on RECIST v1.1
* For Part 1a: Subjects with histologically or cytologically confirmed advanced or metastatic solid tumors that have failed prior standard therapy (including subject refusal or intolerance).
* For Part 1b: Subjects with histologically or cytologically confirmed advanced or metastatic endometrial cancer, gastric cancer, melanoma, microsatellite unstable (MSI) colorectal cancer or other MMR-deficient tumors, non-small cell lung cancer, renal cell carcinoma, head and neck squamous cell carcinoma, triple negative breast cancer, pancreatic ductal carcinoma, or transitional cell carcinoma of the genitourinary tract that have had disease progression after available therapies for advanced or metastatic disease that are known to confer clinical benefit, been intolerant to treatment, or refused standard treatment.
* For Part 1b: Must have documented confirmed disease progression on a prior PD-1 pathway targeted agent or must be PD-1 pathway-targeted treatment naïve.

For Part 2

For subjects with SCLC:

Subjects with histologically or cytologically confirmed advanced or metastatic SCLC. Must not have had previous treatment with antibodies that modulate T-cell function or checkpoint pathways. Must have disease progression on or after platinum-based chemotherapy or must be intolerant to or refuse standard treatment. Must not have received more than 2 lines of prior therapy.

For subjects with NSCLC:

Subjects with a histologically or cytologically confirmed diagnosis of Stage IIIB, Stage IV, or recurrent NSCLC. Have not received more than 1 prior systemic therapy for metastatic NSCLC. No prior therapy with checkpoint inhibitors (anti-PD-1/PD-L1 or anti-CTLA-4). Have confirmation that EGFR or ALK-directed therapy is not indicated as primary therapy (documentation of absence of tumor activating EGFR mutations AND ALK gene rearrangements treatable with a tyrosine kinase inhibitor (TKI) OR presence of a KRAS mutation). If participant's tumor is known to have a predominantly squamous histology, molecular testing for EGFR mutation and ALK translocation will not be required as this is not part of current diagnostic guidelines. Have measurable disease based on RECIST 1.1.

For subjects with UC:

Subjects with a histologically or cytologically confirmed diagnosis of advanced/unresectable (inoperable) or metastatic urothelial cancer of the renal pelvis, ureter, bladder, or urethra. Have had 1 prior treatment of systemic chemotherapy containing a platinum agent or is considered ineligible to receive cisplatin-based combination therapy. No prior therapy with checkpoint inhibitors (anti-PD-1/PD-L1 or anti-CTLA-4). Have measurable disease based on RECIST 1.1.

Exclusion Criteria:

* Laboratory parameters not within the protocol-defined range.
* Receipt of anticancer medications or investigational drugs within a defined interval before the first administration of study drug.
* Received an immune-suppressive based treatment for any reason within 14 days prior to the first dose of study treatment.
* Has not recovered from toxic effect of prior therapy to < Grade 1.
* Active or inactive autoimmune process.
* Has received a live vaccine within 30 days of planned start of study therapy.
* Active infection requiring systemic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 159 (Actual)
Dates: Start 2016-01-25 (Actual); Primary Completion 2019-11-07 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
Part 1: Evaluation of safety and tolerability as measured by the frequency, duration, and severity of adverse events | Duration of study treatment and up to 120 days after the last dose of study drug

SECONDARY OUTCOMES:
Part 1 and 2: Objective Response Rate (ORR) as determined by radiographic disease assessments per immune-related Response Evaluation Criteria In Solid Tumors (irRECIST) v1.1 criteria | Every 9 weeks for the first year on study
Part 1 and 2: Change in the number of Tumor Infiltrating Lymphocytes(TILs) and the ratio of CD8+ lymphocytes to FOXP3+ cells infiltrating tumor post-treatment versus pretreatment by IHC | Up to 5 weeks on study treatment

CONTACTS AND LOCATIONS:
Overall Officials: Peter B. Langmuir, MD, Study Director — Incyte Corporation
Locations (17):
- United States (17):
  - University of California San Francisco Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - John Wayne Cancer Institute at Providence Saint John's Health Center, Santa Monica, California
  - Georgetown University Medical Center Lombardi CCC, Washington D.C., District of Columbia
  - Hematology-Oncology Associates of Treasure Coast, Port Saint Lucie, Florida
  - Emory University, Winship Cancer Institute, Atlanta, Georgia
  - University of Kentucky, Markey Cancer Center, Lexington, Kentucky
  - The Center for Cancer and Blood Disorders (RCCA MD LLC-Maryland Vidision), Bethesda, Maryland
  - Beth Israel Medical Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer institute, Boston, Massachusetts
  - Karmanos Cancer Center, Detroit, Michigan
  - Henry Ford Hospital System, Detroit, Michigan
  - St. Luke's Hospital of Kansas City, Kansas City, Missouri
  - NYU Laura & Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Duke Cancer Institute, Durham, North Carolina
  - UPMC CancerCenters, Hilman Cancer Center, Pittsburgh, Pennsylvania
  - HOPE Cancer Center of East Texas, Tyler, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah

REFERENCES:
- [Derived] Munster P, Iannotti N, Cho DC, Kirkwood JM, Villaruz LC, Gibney GT, Hodi FS, Mettu NB, Jones M, Bowman J, Smith M, Lakshminarayanan M, O'Day S. Combination of Itacitinib or Parsaclisib with Pembrolizumab in Patients with Advanced Solid Tumors: A Phase I Study. Cancer Res Commun. 2023 Dec 19;3(12):2572-2584. doi: 10.1158/2767-9764.CRC-22-0461. PMID 38115208